CLINICAL TRIAL: NCT01465295
Title: Prospective Trial to Evaluate Initial Safety of the HemiBridge™ System in Guided Spinal Growth Treatment of Progressive Idiopathic Scoliosis
Brief Title: Evaluate Initial Safety of the HemiBridge™ System in Guided Spinal Growth Treatment of Progressive Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SpineForm LLC (Industry)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SF001; 11-042 (Other Grant/Funding Number: Ohio Dept of Development Third Frontier Grant); R01FD004144-01 (FDA)
Record Dates: First submitted 2011-10-28; First posted 2011-11-04 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Scoliosis
Keywords: Scoliosis; Adolescent Idiopathic Scoliosis (AIS); Scoliosis treatment; Fusionless spinal surgery; Vertebral stapling; Spinal stapling; Non-fusion; Spinal curvature; Curvature of the spine; Spinal bracing alternative; HemiBridge; SpineForm; Dr. Eric Wall; Dr. George Thompson; Spinal clip; Cincinnati Children's Hospital Medical Center; University Hospitals Case Medical Center, Rainbow Babies
MeSH Terms: conditions — Scoliosis; Spinal Curvatures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HemiBridge (Experimental): Patients meeting eligibility criteria will be treated with the HemiBridge System.
  Interventions: Device: Mechanical hemiepiphysiodesis using the HemiBridge System

INTERVENTIONS:
Device: Mechanical hemiepiphysiodesis using the HemiBridge System — Surgical application of mechanical hemiepiphysiodesis using the HemiBridge device.

SUMMARY:
The purpose of this clinical trial is to study a new method of treatment for patients who are diagnosed with idiopathic scoliosis and have abnormal and increasing curvature of the spine. The treatment consists of the surgical implantation of a new medical device called the "HemiBridge™ Clip". This medical implant device has never been used in humans. SpineForm, LLC, the developer of the HemiBridgeTM System has designed this scientific clinical trial, to evaluate the safety of the use of this device in humans. Information collected from patients treated with this new device shall be used to determine the initial safety of the new device.

The FDA has approved the use of the HemibridgeTM System for this research study in 6 (six) pediatric patients who have idiopathic scoliosis.

This procedure is intended to stop additional curvature of the spine by redirecting growth of the bones of the spine (vertebrae). To accomplish this, the patient undergoes a surgical procedure to securely attach small metal clips (HemiBridge™ Clips) to the outer side of each vertebra involved in the curvature. The HemiBridge™ Clip forms a "bridge" between each vertebra and is intended to hold the vertebrae in place to prevent the spine from curving any further.

DETAILED DESCRIPTION:
Significance Spinal deformity fusion treatment involves some of the most costly and invasive procedures in orthopaedics. The development of an effective treatment method to avoid fusion is needed. Many pediatric spine specialists concur that growth modulation displays compelling pre-clinical and clinical data that must be studied further. While bracing is the only non-operative modality with any evidence of effectiveness for idiopathic scoliosis, its level of effectiveness compared to observation or natural history remains inconclusive. Research has been published for over 50 years, yet conflicting literature reports both successes and failures. Most literature consists of retrospective reports of bracing experience, with little commonality relative to existing conditions at the time bracing is initiated, documentation of compliance and basis for judging success.

The U.S. Preventative Services Task Force (USPSTF) is an independent panel of private-sector experts in primary care and prevention. The Task Force was convened by the U.S. Public Health Service to systematically review the evidence of effectiveness of clinical preventive services. One of their charges was to evaluate the evidence supporting the practice of school screening for adolescent idiopathic scoliosis. After systematically reviewing the literature to date, their policy statement issues in 1992, and updated in 1996 states "…There is inadequate evidence to determine whether brace therapy limits the natural progression of the disease in a significant proportion of cases, as most studies suffer from selection bias, lack of internal control groups, inadequate follow-up, small sample sizes, and lack of health outcome measures."

There is no Level One evidence to support the practice of bracing, and clinicians are left with conflicting and questionable inferences regarding bracing effectiveness. Some clinicians believe the evidence favors a decrease in the rate of curve progression, and based on this assumption, over half the states in the U.S. have mandated school screening programs for the detection and early treatment of scoliosis. On the other hand, groups such as the USPSTF, its British and Canadian counterparts and many individual practitioners worldwide feel the evidence is inconclusive and are therefore ambivalent about brace treatment.

Due to the variability in published results on brace effectiveness, researchers in the United States and Canada have commenced a randomized multi-center trial of bracing versus no bracing to determine the effectiveness of brace wear in the treatment of idiopathic scoliosis (BRAIST Study). This study, which was initiated in 2007 in the United States, is being performed under the auspices of the US National Institutes of Health (NIH) and Canadian Institute of Health. In the Netherlands, a randomized multi-center study comparing bracing to observation is also underway.

While bracing treatment is non-invasive and preserves growth, motion and function of the spine, it does not correct the deformity. In addition, the brace pressure on the rib cage and the influence on the chest wall in a growing child create concerns. Some scoliosis patients wear a brace for as long as five years only to learn that brace treatment failed and then recommended to endure major fusion surgery and recovery.

When surgery (fusion and instrumentation) is required for scoliosis, internal fixation of the spine to achieve correction and bony fusion is performed. Surgical correction via posterior fusion is typically performed for curves greater than 40 - 50°, often with accompanying discectomy and release of the anterior longitudinal ligaments for curves greater than 75°. Smaller incisions or use of portals for anterior surgery became available in the early 1990's with video-assisted thoracoscopic surgery (VATS). Potential advantages include less muscular and chest wall disruption, less impact on pulmonary function, quicker recovery time and smaller scars. Arlet (2000) completed a meta-analysis of 10 articles with a total of 151 patients, where VATS was utilized in scoliosis surgery. Of the 151 patients, 18% (27 complications) experienced major and minor complications, including major bleeding (3), prolonged ventilation (10), pulmonary complications (6), intercostal neuralgia (number not specified), aborted procedure (3), and one each chylothorax, infection, and tachycardia. A conclusion could not be drawn as to whether the complication rate is increased or decreased with VATS. The correction rate was similar to open thoracotomy.

Scoliosis fusion surgery involves extensive posterior and/or anterior spine exposure with associated risks, frequent blood transfusions (2 to 4 units), high postoperative pain, loss of motion of the treated segment, and slow rehabilitation. The child also has potential life-long complications that do not present for several years after surgery, including adjacent segment disease or degeneration that in many cases requires additional surgery.

Andersen conducted a study of 100 braced and 115 surgical patients with idiopathic scoliosis 10 years after the treatment was completed. The SF-36 scores (patient physical and mental health assessment) did not differ between the two groups; however, both group's scores were lower than age-matched normal controls. Results for the braced patients indicated that 17% felt that the brace was so unpleasant that they would rather take the chance of curve progression than wear a brace. Of the braced patients, 71% indicated that they would have preferred an operation (fusion) to a brace. More than two of three patients didn't wear the brace as prescribed due to skin irritation. Other investigators have refuted the impact of bracing on the quality of life.

Thus, neither bracing nor surgical fusion treatments represent an ideal treatment of idiopathic scoliosis. As such, there is a need for idiopathic scoliosis treatments that address the population of patients whose curvature is unlikely to be corrected via bracing but for whom the risks of less invasive non-fusion surgical treatment may be exceeded by the potential benefit in avoiding lifelong progression or an extensive fusion surgery.

The HemiBridge™ System is indicated for progressive idiopathic scoliosis (Lenke Type 1A or 1B) in skeletally immature (Risser Grade 0 and triradiate cartilage open) patients by mechanically modulating spinal growth (hemiepiphysiodesis) and arresting spinal deformity progression without the need for spinal fusion. The HemiBridge™ System is intended to be placed at contiguous levels through an anterior thoracoscopic procedure on the convex side of a main thoracic curve that measures 25° to 40°, where the end of the vertebrae of the curve spans levels inclusive of or between T3 and L1. The HemiBridge™ System is intended for males and females with a chronologic age of 10 years and older. Females with an Atlas Matching bone age ≥ 8 years and 10 months not to exceed 13 years (or pre-menarche) and males with an Atlas Matching bone age ≥ 10 years not to exceed 15 years.

Innovation The study device, named the HemiBridgeTM System, is the result of extensive pre-clinical research and development initiated by Donita Bylski-Austrow, PhD and Eric Wall, MD both of Cincinnati Children's Hospital Medical Center and the University of Cincinnati. Research and development of the study device to date has used an interdisciplinary team, including pediatric spine surgeons, engineers, scientists and regulatory experts. This team has helped define the compressive loading required to alter growth, tested prototype devices in preclinical models, improved the test articles for clinical use, and confirmed repeatable in-vivo results in compliance with FDA Good Laboratory Practices. This process has led to the approval of a study device that has achieved FDA and IRB approvals to begin clinical phase testing.

The HemiBridge System's innovation is in its ability to apply mechanical hemiepiphysiodesis to redirect spine growth and developed to accommodate adolescent physiologic loading while remaining securely fastened to the spinal motion segment. Additionally, the System includes innovative patient safety and surgeon interface features. The surgical technique and instrumentation were co-developed by SpineForm LLC and the Orthopaedics Department at Cincinnati Children's Hospital Medical Center.

The application of mechanical hemiepiphysiodesis to treat progressive scoliosis challenges the use of external bracing and/or observation (watchful waiting). Comparing the pooled rates for these two non-operative interventions shows no clear advantage of either approach; therefore, one cannot recommend one non-operative approach over the other to prevent the need for surgery in adolescent idiopathic scoliosis. Arresting curve progression with the HemiBridge System and avoiding fusion may significantly impact quality of life while reducing total lifetime patient care cost. Providing patients with a surgical alternative that is superior to the current non-operative standard of care is a paradigm shift that must be studied further to determine its safety and indications for use.

The clinical study protocol design is limited to patients at the highest risk of progressing to needing multi-level fusion surgery. There are no medical devices cleared by the FDA to treat late juvenile or early adolescent onset of idiopathic scoliosis. The HemiBridge System is the first mechanical compression device FDA approved for pediatric investigational use. The proposed study is the first use in humans of the HemiBridge System. The clinical trials will enable the study sponsor to gather prospective information to continuously improve the product, its indications, the next study phase clinical protocol design and recommended surgical technique.

ELIGIBILITY:
Inclusion Criteria:

- Patients must meet all the criteria to be enrolled in this study:

* Trial subject population will involve patients who are skeletally immature, who have a diagnosis of idiopathic scoliosis with a single main thoracic curve Cobb angle 25° to 40° and Lenke Type 1A or 1B.

  1. Chronologic age:

     * Males ≥ 10 years
     * Females ≥ 10 years
  2. Females pre-menarchal at screening examination
  3. Bone age as confirmed by radiographs of left hand and wrist according to the "Atlas Matching" method of Greulich and Pyle:

     * Females: ≥ 8 years and 10 months not to exceed 13 years
     * Males: ≥ 10 years not to exceed 15 years
  4. Skeletal immaturity (Risser grade 0 and the triradiate cartilage is open) as determined by standing, upright PA radiograph. If radiographic Risser grade results are indeterminate, the bone age from the Atlas Matching will prevail.
  5. Main thoracic Cobb angle of 25° to 40° as determined from standing, upright PA radiographs where the end vertebra are between or including T3 and L1 without wearing a brace
  6. Clinical diagnosis of idiopathic scoliosis with a single main thoracic curve as determined with measurement on standing posterior- anterior PA radiographs.

     * Defined as a single thoracic curve where either: central sacral vertical line (CSVL) passes between the pedicles of the apical lumbar vertebra; or the CSVL touches the lumbar apical body(ies) (Lenke Type 1A or 1B, respectively)
  7. Achievable anatomical fit as determined by calibrated standing PA film:

     * Disc height not exceeding 10 mm at each spinal level to be instrumented relative to location of the probable implant and
     * Minimum central vertebral height that will accept the selected HemiBridge™ Clip size at all levels planned for implants
  8. BMI < 30
  9. Physical and mental ability to undergo surgery with single lung ventilation
  10. Written informed assent from the patient
  11. Written informed consent from parent and/or legal guardian and authorization to use protected health information (by Sponsor, third party core lab and/or clinical evaluation committee)

Exclusion Criteria:

* Patients who meet any of the exclusion criteria will not be enrolled.

  1. Non-idiopathic scoliosis
  2. Males and females chronological age < 10 years
  3. Triradiate cartilage is closed as determined on the standing PA radiograph at baseline screening
  4. Any curve type that does not meet definition of Lenke 1A or 1B
  5. Any main thoracic deformity that measures < 25° or > 40° Cobb angle
  6. Any main thoracic deformity that includes vertebral levels including and cranial to T2
  7. Any main thoracic deformity that includes vertebral levels including and caudal to L2
  8. Prior thoracotomy, thoracostomy or any spine surgery
  9. T3-T12 kyphosis > 40° (T4 or T5-T12 if visualization impaired at T3)
  10. Known history or existing malignancy, or any systemic or local infection
  11. Spinal cord abnormalities that require treatment
  12. Presence of neurological deficit (motor grades 0-4, sensory grades 0-1, reflexes grade 0 or 5 or asymmetry of deep tendon reflexes > 2 from right to left)
  13. Insulin-dependent diabetes
  14. Severe asthma
  15. Reduced pulmonary function, defined as < 60% of predicted value (Forced expiratory volume in one second [FEV1] divided by forced vital capacity [FVC]) or Subject has moderately severe or worse ventilatory limitation defined as < 60% of predicted value of the forced vital capacity [FVC] for age, race, sex and height (with height determined by arm span in patients with scoliosis and reference equations derived from the data of Wang et al 199329.)
  16. Cardiopulmonary or other systemic disease
  17. Bleeding disorder(s)
  18. Ataxia
  19. Documented HIV or hepatitis infection
  20. Family history of neurofibromatosis or Marfan's syndrome
  21. Medical contraindication to anesthesia
  22. Suspected or known allergy to titanium
  23. Not available for interval visits and long term follow-up exams

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-08; Primary Completion 2017-12-29 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
Acute Safety: Incidence, relatedness (relationship to procedure and device), seriousness and severity of Adverse Events By Participant | 1 month post-operative
  Incidence, relatedness (relationship to procedure and device), seriousness and severity of Adverse Events By Participant

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E Reynolds, MBA, Study Director — SpineForm LLC; Eric J Wall, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Case Medical Center - Rainbow Babies & Children's Hospital, Cleveland, Ohio

REFERENCES:
- [Background] Bunge EM, de Koning HJ; brace trial group. Bracing patients with idiopathic scoliosis: design of the Dutch randomized controlled treatment trial. BMC Musculoskelet Disord. 2008 Apr 22;9:57. doi: 10.1186/1471-2474-9-57. PMID 18430217
- [Background] Guille JT, D'Andrea LP, Betz RR. Fusionless treatment of scoliosis. Orthop Clin North Am. 2007 Oct;38(4):541-5, vii. doi: 10.1016/j.ocl.2007.07.003. PMID 17945133
- [Background] Wiggins GC, Shaffrey CI, Abel MF, Menezes AH. Pediatric spinal deformities. Neurosurg Focus. 2003 Jan 15;14(1):e3. doi: 10.3171/foc.2003.14.1.4. PMID 15766220
- [Background] Lonner BS. Emerging minimally invasive technologies for the management of scoliosis. Orthop Clin North Am. 2007 Jul;38(3):431-40; abstract vii-viii. doi: 10.1016/j.ocl.2007.03.011. PMID 17629990
- [Background] Arlet V. Anterior thoracoscopic spine release in deformity surgery: a meta-analysis and review. Eur Spine J. 2000 Feb;9 Suppl 1(Suppl 1):S17-23. doi: 10.1007/s005860000186. PMID 10766053
- [Background] Vaccaro AR, Regan JJ, Crawford AH, Benzel EC, Anderson DG. Complications of pediatric and adult spinal surgery. Chapter 7, Postarthrodesis Adjacent Segment Degeneration, Marcel Dekker, New York, 2004; p 82.
- [Background] Andersen MO, Christensen SB, Thomsen K. Outcome at 10 years after treatment for adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2006 Feb 1;31(3):350-4. doi: 10.1097/01.brs.0000197649.29712.de. PMID 16449910
- [Background] Dolan LA, Weinstein SL. Surgical rates after observation and bracing for adolescent idiopathic scoliosis: an evidence-based review. Spine (Phila Pa 1976). 2007 Sep 1;32(19 Suppl):S91-S100. doi: 10.1097/BRS.0b013e318134ead9. PMID 17728687
- [Background] Bylski-Austrow DI, Wall EJ, Rupert MP, Roy DR, Crawford AH. Growth plate forces in the adolescent human knee: a radiographic and mechanical study of epiphyseal staples. J Pediatr Orthop. 2001 Nov-Dec;21(6):817-23. PMID 11675562
- [Background] Wall EJ, Bylski-Austrow DI, Kolata RJ, Crawford AH. Endoscopic mechanical spinal hemiepiphysiodesis modifies spine growth. Spine (Phila Pa 1976). 2005 May 15;30(10):1148-53. doi: 10.1097/01.brs.0000162278.68000.91. PMID 15897828
- [Background] Bylski-Austrow DI, Wall EJ, Glos DL, Ballard ET, Montgomery A, Crawford AH. Spinal hemiepiphysiodesis decreases the size of vertebral growth plate hypertrophic zone and cells. J Bone Joint Surg Am. 2009 Mar 1;91(3):584-93. doi: 10.2106/JBJS.G.01256. PMID 19255218
- [Derived] Wall EJ, Reynolds JE, Jain VV, Bylski-Austrow DI, Thompson GH, Samuels PJ, Barnett SJ, Crawford AH. Spine Growth Modulation in Early Adolescent Idiopathic Scoliosis: Two-Year Results of Prospective US FDA IDE Pilot Clinical Safety Study of Titanium Clip-Screw Implant. Spine Deform. 2017 Sep;5(5):314-324. doi: 10.1016/j.jspd.2017.02.004. PMID 28882349
- See also: Website to contact SpineForm LLC — http://spineform.com